CLINICAL TRIAL: NCT03232905
Title: A Phase 1, Randomized, Double-blind, Third-party Open, Placebo-controlled Study To Evaluate The Safety, Tolerability, And Pharmacokinetics After Multiple Oral Doses Of Pf-06651600 In Healthy Japanese Subjects
Brief Title: Safety and Pharmacokinetic Study of PF-06651600 in Japanese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B7981008; 2017-001298-17 (EudraCT Number)
Record Dates: First submitted 2017-07-25; First posted 2017-07-28 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Healthy
MeSH Terms: interventions — PF-06651600

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PF-06651600 (Experimental): Multiple ascending doses of PF-06651600
  Interventions: Drug: PF-06651600
- Placebo (Placebo Comparator): Multiple ascending doses of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06651600 — PF-06651600 will be administered as tablet
  Arms: PF-06651600
Drug: Placebo — Matching placebo will be administered as tablet
  Arms: Placebo

SUMMARY:
This study is a phase 1 study of PF-06651600. PF-06651600 is being developed for treatment of inflammatory bowel disease. The goal of the study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of PF-06651600 after multiple oral doses of PF-06651600 in Japanese healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have four Japanese grandparents who were born in Japan.
* Healthy male subjects and/or female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive
* No evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB)
* BMI of 17.5 to 27.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Evidence of personally signed and dated informed consent document.
* Willing and able to comply with scheduled visits, treatment plan, lab tests and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, GI, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* Males of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product
* Use of tobacco/nicotine containing products in excess of 5 cigarettes/day.
* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males.
* Screening blood pressure >140/90 mm Hg.
* Screening laboratory abnormalities as defined by the protocol.
* Unwilling or unable to comply with the Lifestyle Guidelines as defined by the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-11-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (AEs), Serious Adverse Events (SAEs) and Discontinuation Due to AEs | Baseline up to Day 45
Change From Baseline in 12-Lead Electrocardiogram (ECG) Parameters (PR Interval, QRS interval, QT Interval, QTC Interval, heart rate) | Baseline, 1 hour post-dose on Day 1 and 10
Change From Baseline in Vital Signs (Blood Pressure, Pulse Rate, Oral Temperature) | Baseline, Day 1, 10, 12 and 28
Number of Participants With Change From Baseline in Physical Examinations | Baseline up to Day 28
Number of Participants With Laboratory Abnormalities | Baseline up to Day 28

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of PF-06651600 at Day 1 | pre-dose 0.5, 1, 2, 4, 6, 8, 12, 16, 24 hour post-dose on Day 1
Maximum Observed Plasma Concentration (Cmax) of PF-06651600 at Day 10 | pre-dose 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hour post-dose on Day 10
Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06651600 at Day 1 | pre-dose 0.5, 1, 2, 4, 6, 8, 12, 16, 24 hour post-dose on Day 1
Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06651600 at Day 10 | pre-dose 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hour post-dose on Day 10
Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinite Time (AUCinf) of PF-06651600 at Day 1 | pre-dose 0.5, 1, 2, 4, 6, 8, 12, 16, 24 hour post-dose on Day 1
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-06651600 at Day 1 | pre-dose 0.5, 1, 2, 4, 6, 8, 12, 16, 24 hour post-dose on Day 1
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-06651600 at Day 1 | pre-dose 0.5, 1, 2, 4, 6, 8, 12, 16, 24 hour post-dose on Day 1
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-06651600 at Day 10 | pre-dose 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hour post-dose on Day 10
Plasma Decay Half-Life (t1/2) of PF-06651600 at Day 1 | pre-dose 0.5, 1, 2, 4, 6, 8, 12, 16, 24 hour post-dose on Day 1
Plasma Decay Half-Life (t1/2) of PF-06651600 at Day 10 | pre-dose 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hour post-dose on Day 10
Observed Accumulation Ratio (Rac) on AUCtau for PF-06651600 at Day 10 | pre-dose 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hour post-dose on Day 10
Observed Accumulation Ratio on Cmax (RacCmax) for PF-06651600 at Day 10 | pre-dose 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hour post-dose on Day 10
MinimumObserved Plasma Concentration (Cmin) of PF-06651600 at Day 10 | pre-dose 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hour post-dose on Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Wojciechowski J, S Purohit V, Huh Y, Banfield C, Nicholas T. Evolution of Ritlecitinib Population Pharmacokinetic Models During Clinical Drug Development. Clin Pharmacokinet. 2023 Dec;62(12):1765-1779. doi: 10.1007/s40262-023-01318-3. Epub 2023 Nov 2. PMID 37917289
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7981008&StudyName=A+Phase+1%2C+Randomized%2C+Double-blind%2C+Third-party+Open%2C+Placebo-controlled+Study+To+Evaluate+The+Safety%2C+Tolerability%2C+And+Pharmacokinetics+After+Multiple+Oral+Doses+Of+Pf-06651600+In+Healthy+Japanese+Subjects